CLINICAL TRIAL: NCT01660295
Title: An Open-label, Single Center, Parallel-group Study to Compare the Single- and Repeated-dose Pharmacokinetics of Stepwise Increasing Doses of Subcutaneous Certoparin (3000 IU o.d., 3000 IU b.i.d., 8000 IU o.d., and 8000 IU b.i.d.) in Subjects With Severe Renal Insufficiency and Healthy Subjects
Brief Title: Pharmacokinetics of Certoparin in Subjects With Renal Insufficiency and Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMEX839BDE07; 2011-001930-40 (EudraCT Number)
Record Dates: First submitted 2011-12-20; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Renal Insufficiency
Keywords: Severe renal insufficiency certoparin; Severe renal insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — certoparin

ARMS (2):
- Certoparin control (Experimental): Participants receive Certoparin 3,000 IU during period 1. Participants will receive 8,000 IU during period 2, if qualified as per medical criteria.
  Interventions: Drug: Certoparin 3,000 IU Once Daily; Drug: Certoparin 8,000 IU Twice a Day
- Certoparin Renal (Experimental): Participants receive dose escalation upon medical criteria qualification at each period:
  Certoparin 3,000 IU once a day during period 1. Certoparin 3,000 IU twice a day during period 2. Certoparin 8,000 IU once a day during period 3. Certoparin 8,000 IU in the morning and 3,000 IU in the evening during period 4 OR Certoparin 8,000 IU twice a day during period 4.
  Interventions: Drug: Certoparin 3,000 IU Once Daily; Drug: Certoparin 3,000 IU Twice a Day; Drug: Certoparin 8,000 IU Once Daily; Drug: Certoparin 8,000 IU Twice a Day

INTERVENTIONS:
Drug: Certoparin 3,000 IU Once Daily — Certoparin 3,000 IU subcutaneous injection once daily
  Other Names: Mono-Embolex
Drug: Certoparin 3,000 IU Twice a Day — Certoparin 3,000 IU subcutaneous injection twice a day
  Other Names: Mono-Embolex
  Arms: Certoparin Renal
Drug: Certoparin 8,000 IU Once Daily — Certoparin 8,000 IU subcutaneous injection once daily
  Other Names: Mono-Embolex
  Arms: Certoparin Renal
Drug: Certoparin 8,000 IU Twice a Day — Certoparin 8,000 IU subcutaneous injection twice a day
  Other Names: Mono-Embolex

SUMMARY:
This study will assess the pharmacokinetics in subjects with severe renal insufficiency and healthy subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects OR
* Subjects with severe renal insufficiency

Exclusion criteria:

* Hypersensitivity to study medication
* Genetic abnormality or disease of clotting system
* Prior major surgery or bleeding
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Plasma aXa-Profile: C0 | 5 days
  Estimate of the effects of renal insufficiency on the systemic exposure to aXa for once daily (τ = 24 h) repeated doses of 3,000 IU aXa as characterized by pre-dose trough (C0,ss) aXa comparing REN-patients with matched CON-subjects studied in parallel.
Dose regimen, systemic total exposure to aXa (AUC0-τ,ss) | 5 days
  Dosage regimen (3,000 o.d., 3,000 b.i.d., 8,000 o.d., 8,000 IU aXa in the morning plus 3,000 IU aXa in the evening, or 8,000 b.i.d. IU aXa) that yields a systemic total exposure to aXa (AUC0-τ,ss) in REN-patients similar to that achieved with 8,000 b.i.d. IU aXa in CON-subjects.
Plasma aXa-Profile: Cmax | 5 days
  Estimate of the effects of renal insufficiency on the systemic exposure to aXa for once daily (τ = 24 h) repeated doses of 3,000 IU aXa as characterized by maximum (Cmax,ss), aXa comparing REN-patients with matched CON-subjects studied in parallel.
Plasma aXa-Profile: AUC | 5 days
  Estimate of the effects of renal insufficiency on the systemic exposure to aXa for once daily (τ = 24 h) repeated doses of 3,000 IU aXa as characterized by total (AUC0-τ,ss) aXa comparing REN-patients with matched CON-subjects studied in parallel.

CONTACTS AND LOCATIONS:
Locations (1):
- DRC Drug Research Center Ltd., H-8230 Balatonfüred, H-8230 Balatonfüred, Ady E. U., Hungary